CLINICAL TRIAL: NCT05222100
Title: Effect of Breast Implants om Mammography Screening
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-01534
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; plastic surgery; breast implant; mammography screening; health economy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women without breast implants: Women without breast implants participating in the mammography screening program.
  Interventions: Diagnostic Test: Mammography screening
- Women with breast implants: Women with breast implants participating in the mammography screening program.
  Interventions: Diagnostic Test: Mammography screening

INTERVENTIONS:
Diagnostic Test: Mammography screening — Breast screening mammograms use X-rays to look for cancers that are too small to see or feel.
  Other Names: Mammogram screening; Breast screening; Screening mammogram; Screening mammography; Breast cancer screening

SUMMARY:
The purpose of the study is to survey how many women have breast implants in the mammography screening population and the effect of implants on the number and type of examinations and on costs.

ELIGIBILITY:
Inclusion Criteria:

* Women participating in the mammography screening program.

Exclusion Criteria:

* None

Ages: 40 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological women included in the mammography screening program.
Study Population: Women participating in the mammography screening program in Gothenburg, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Costs | 1 year post-operatively
  Health economic analysis of the effects of implants on mammography screening

SECONDARY OUTCOMES:
Prevalence | 1 year
  Prevalence of breast implants in a mammography screening population.
Frequency of need for additional examinations | 1 year
  Survey of if breast implants infer extra examinations (mammography, ultrasounds, biopsies, diagnostic operations) in connection with screening mammography.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansson E, Zaya S, Meyer S, Freiin von Wrangel A, Warnberg F, Zackrisson S. Prevalence of women with breast implants in Sweden: a study based on the population-based mammography screening programme. J Plast Surg Hand Surg. 2023 Sep 20;58:96-100. doi: 10.2340/jphs.v58.15298. PMID 37728392
- See also: Research group — https://www.gu.se/forskning/rekonstruktiv-brostkirurgi